CLINICAL TRIAL: NCT04848350
Title: The Effect of Inhaler Lavender and Frankincense Aromatherapy on Pain and Anxiety in Patients Undergoing SWL.
Brief Title: Use of Inhaler Aromatherapy During SWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Barıs Saylam, M.D., Mersin Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020376
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Pain, Procedural; Aromatherapy; Anxiety
Keywords: aromatherapy; lavender; frankincense
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders | interventions — lavender oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo group (Placebo Comparator): Only a saline solution was applied to the placebo group
  Interventions: Other: Lavender essential oil
- lavender group (Active Comparator): The lavender essential oil was added to the nebulizer and operated on in the SWL room before the procedure,
  Interventions: Other: Lavender essential oil
- frankincense group (Active Comparator): The frankincense essential oil was added to the nebulizer and operated on in the SWL room before the procedure,
  Interventions: Other: Lavender essential oil

INTERVENTIONS:
Other: Lavender essential oil — Aromatherapy agents were added to the nebulizer at a rate of 2% (120 ml of water).The nebulizer was prepared and operated on in the SWL room before the procedure, The patients were taken to the room 5 minutes before the procedure and the nebulizer was operated on during the procedure
  Other Names: frankincense essential oil

SUMMARY:
The study aims to determine the effects of inhalation aromatherapy on pain and anxiety during the SWL protocol. This study included 120 patients who were scheduled to undergo SWL. Patients were randomly assigned a control placebo group 1 (n=40), the lavender group 2 (n=40), and the frankincense group 3 (n=40). The nebulizer (a rate of 2%) was prepared and operated on in the SWL room before the procedure. Data were collected using the visual analog scale (VAS) and the State Anxiety Inventory (STAI-I).

DETAILED DESCRIPTION:
Shock Wave Lithotripsy (SWL) is widely and effectively used in the treatment of urinary tract stone disease. In the first applied lithotriptors, the energy density and maximum energy application at the skin level revealed the need for anesthesia in terms of pain. Later, with the development of new devices, the physics parameters were changed and shock was applied with lower energy levels, using large ellipsoids, the area where shock waves enter the skin is reduced and anesthesia is restricted. During the SWL procedure, patients can identify pain in the form of a subjective sensation that is difficult to identify. Pain occurs for two reasons. The first is the trauma caused by shock waves moving towards the kidney as they pass through the skin and muscles, and the second is the deep organ pain due to the trauma caused by shock waves in the kidney Also, various patient-related and environmental factors affecting pain should be considered. The sedation of patients greatly facilitates SWL tolerance. However, it has been noted in various studies that patients with anxiety experience more pain during SWL. Aromatherapy is a TAT (Tapas Acupressure technique) method in which essential oils created from fragrant parts of plants are absorbed from the body and show their effects. The therapeutic, disease-relieving or preventive properties of essential oils are utilized. Essential oils can be applied to the body by topical, internal, oral, and inhalation methods. The fastest and easiest way of entry of essential oils into the body is inhalation. When applied through breathing, evaporating molecules reach the olfactory bulb through the nose and the limbic system in the brain. Aromatherapy provides control of pain and anxiety by affecting the amygdala and hippocampus, which regulate fear and aggressive behaviors in the limbic system. Aromatherapy by Inhaler is used in hemodialysis, dental procedures, intrauterine contraceptive placement, pain and anxiety control in patients with arthritis. The literature shows that Lavender (lavandula officinalis) and Frankincense (Boswellia) essential oils are used in pain and anxiety management in procedural pain and anxiety control.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing SWL
* Ages between 18-60

Exclusion Criteria:

* Patients with pain before the procedure (VAS value is non-zero)
* Patients with respiratory disease (lung cancer, asthma, bronchitis, chronic obstructive pulmonary disease, etc.),
* patients using painkillers in the last 3 hours,
* patients who were disturbed by the smell of used essential oils
* patients with a known allergy to used essential oils with a history of contact dermatitis against cosmetic odor.
* Patients who used anxiolytic agents and narcotics were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
VAS score | 10 minutes
  Patients ' pain levels were measured using the VAS pain scale. This is a horizontal scale, ranging from 0 (no pain) on the left side to 10 (most severe pain) on the right side. Pain intensity can be categorized as mild (score, 1-3), moderate (score, 4-6), and severe (score, 7-10) according to the scale.
Discomfort Intolerance Scale-Revised (DIS-R) | 10 minutes
  The scala assesses the perceived inability to tolerate physical discomfort, beliefs about physical discomfort, and responses to feelings of physical discomfort. The DIS-R consists of nine items (e.g., "I can't handle feeling physical discomfort") rated on a 7-point Likert-type scale (0=not at all like me to 6=extremely like me) with higher scores indicating greater discomfort intolerance. Confirmatory factor analysis revealed that the revised 9-item version was a good fit to the data and demonstrated good construct validity in both symptomatic (i.e., clinically-elevated levels of depression or anxiety) and non-symptomatic samples.
STAI form | 10 minutes
  The STAI form was used to determine the transitory emotional state and anxiety level of the participants after the procedure. This scale, consisting of 20 items, uses a 4-point Likert scale in which items are scored from 1 (not at all) to 4 (very much). The assessment of the inventory is based on the total score ranging from 20 to 80. A score from1 to 20 is considered to indicate no anxiety, a score of 21 to 40 indicates mild anxiety, a score of 41 to 60 indicates moderate anxiety, and a score of 61 and higher indicates severe anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Erim Erdem, Prof., Principal Investigator — Mersin University Scholl of Medicine
Locations (1):
- Barış Saylam, Mersin, Mezitli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barati F, Nasiri A, Akbari N, Sharifzadeh G. The Effect of Aromatherapy on Anxiety in Patients. Nephrourol Mon. 2016 Jul 31;8(5):e38347. doi: 10.5812/numonthly.38347. eCollection 2016 Sep. PMID 27878109
- [Background] Cai H, Xi P, Zhong L, Chen J, Liang X. Efficacy of aromatherapy on dental anxiety: A systematic review of randomised and quasi-randomised controlled trials. Oral Dis. 2021 May;27(4):829-847. doi: 10.1111/odi.13346. Epub 2020 May 26. PMID 32267044
- [Background] Tabatabaeichehr M, Mortazavi H. The Effectiveness of Aromatherapy in the Management of Labor Pain and Anxiety: A Systematic Review. Ethiop J Health Sci. 2020 May;30(3):449-458. doi: 10.4314/ejhs.v30i3.16. PMID 32874088
- [Result] Jaruzel CB, Gregoski M, Mueller M, Faircloth A, Kelechi T. Aromatherapy for Preoperative Anxiety: A Pilot Study. J Perianesth Nurs. 2019 Apr;34(2):259-264. doi: 10.1016/j.jopan.2018.05.007. Epub 2018 Sep 8. PMID 30205934
- [Result] Ozkaraman A, Dugum O, Ozen Yilmaz H, Usta Yesilbalkan O. Aromatherapy: The Effect of Lavender on Anxiety and Sleep Quality in Patients Treated With Chemotherapy. Clin J Oncol Nurs. 2018 Apr 1;22(2):203-210. doi: 10.1188/18.CJON.203-210. PMID 29547610
- [Result] Gong M, Dong H, Tang Y, Huang W, Lu F. Effects of aromatherapy on anxiety: A meta-analysis of randomized controlled trials. J Affect Disord. 2020 Sep 1;274:1028-1040. doi: 10.1016/j.jad.2020.05.118. Epub 2020 May 26. PMID 32663929